CLINICAL TRIAL: NCT01428596
Title: A Phase I Dose-escalation Clinical Trial to Evaluate the Safety and Immunogenicity of a Replication-defective HIV-1 Vaccine (HIVAX™) in HIV-1 Infected Subjects Receiving Highly Active Antiretroviral Therapy
Brief Title: Safety and Immunogenicity of HIVAX in HIV-1 Infected Subjects
Acronym: GCHT01
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GeneCure Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A010
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: HIV Infections
Keywords: HIV-1; therapeutic vaccine; immunotherapy; AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Experimental): Lower dose HIVAX vaccine
  Interventions: Biological: HIVAX
- Arm II (Placebo Comparator): lower dose, placebo control
  Interventions: Biological: saline solution
- Arm III (Experimental): Higher dose HIVAX vaccine
  Interventions: Biological: HIVAX

INTERVENTIONS:
Biological: HIVAX — Vaccine 1.0 ml SQ lower dose (10^8 TU) at weeks 0, 8 and 16.
  Arms: Arm I
Biological: saline solution — Saline solution 1.0 ml SQ at weeks 0, 8 and 16.
  Arms: Arm II
Biological: HIVAX — Vaccine 1.0 ml SQ higher dose (10^9 TU) at weeks 0, 8 and 16.
  Arms: Arm III

SUMMARY:
This study is to test a therapeutic HIV-1 vaccine (HIVAX™) in HIV-1 infected subjects. The safety and immune responses will be studied in vaccine recipients. The anti-viral effect of HIVAX vaccine will be monitored during a 12-week treatment interruption phase.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled dose-escalation clinical trial to evaluate the safety and the immunogenicity of two doses of a replication defective HIV-1 vaccine (HIVAX™) in subjects receiving stable highly active antiretroviral therapy (HAART) who have an HIV-1 RNA <50 copies/ml and CD4 cell count >500 cells/mm3. Following the randomized placebo-controlled vaccination phase subjects who received active vaccine and who meet eligibility will undergo a 12-week analytical antiretroviral treatment interruption followed by reinstitution of antiretroviral therapy (or continued interruption) with follow up through week 48.

ELIGIBILITY:
Part I (vaccination phase) Inclusion Criteria:

1. HIV-1 infection, as documented by any licensed ELISA test kit and confirmed by Western blot, at any time prior to study entry. HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
2. On highly active antiretroviral therapy defined as the combination of at least three antiretroviral agents for at least 12 months prior to study entry.

   NOTE: A regimen that included only the combination of 3 NRTIs alone will not meet the study definition of a highly active antiretroviral therapy regimen. The combination of low dose ritonavir and another PI will be considered as one antiretroviral agent. Subjects cannot be on an NNRTI containing regimen at study entry.
3. Subjects must be on a stable regimen (no change in therapy) for at least 2 months prior to study entry.

   NOTE: A change in formulation or class for reasons other than virologic failure will be allowed but must have documented viral suppression (HIV RNA <50 copies/ml) on at least two consecutive measurements at least two weeks apart.
4. Prior sustained response to antiretroviral therapy defined as an HIV-1 RNA <50 copies/ml and a CD4 cell count >500 cells/mm3 for twelve months prior to study entry documented on at least three measurements prior to study entry.

   NOTE: cannot have any confirmed HIV-1 RNA ≥50 copies/ml during the 12-months prior to study entry.
5. CD4 cell count >500 cells/mm3 within 60 days prior to study entry at any laboratory that has a CLIA certification or its equivalent.
6. HIV-1 RNA <50 copies/ml obtained within 30 days prior to study entry by any laboratory that has a CLIA certification or its equivalent.
7. Willingness to interrupt all antiretroviral therapy for at least 12 weeks following completion of vaccination phase (Part I).
8. Laboratory values obtained within 30 days prior to study entry.

   * Absolute neutrophil count (ANC) ≥ 750/mm3.
   * Hemoglobin ≥ 8.5 g/dL.
   * Platelet count ≥ 75,000/mm3.
   * AST (SGOT), ALT (SGPT), and alkaline phosphatase ≤ 2.5 x ULN.
   * Total bilirubin ≤ 2.5 x ULN.
   * PT < 1.2 ULN and PTT < 1.5 ULN NOTE: Asymptomatic subjects with total bilirubin ≥2.5 x ULN, receiving indinavir and/or atazanavir are eligible.
9. Negative pregnancy test within 14 days prior to study entry.
10. Willingness to use adequate contraception by study participants

    Subjects must agree not to participate in a conception process (e.g., active attempts to become pregnant or to impregnate, sperm donation, or in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, subjects must use a form of contraception as listed below while on study vaccine and for 60 days after stopping study vaccine.

    Women without reproductive potential (i.e., have reached menopause or undergone hysterectomy, bilateral oophorectomy, or tubal ligation) or women whose male partner has undergone successful vasectomy with documented azoospermia or has documented azoospermia for any other reason, are eligible without requiring the use of contraception.

    NOTE: Subject-reported history is acceptable documentation of sterilization (hysterectomy, bilateral oophorectomy, tubal ligation, or vasectomy).

    As appropriate, at least one of the following methods must be used appropriately with or without a hormonal-based method during the study:
    * Condoms (male or female) with or without a spermicidal agent.
    * Diaphragm or cervical cap with spermicidal agent
    * IUD
11. Karnovsky performance score ≥ 90.
12. Men and women ≥ 18 years of age and < 60 years of age.
13. Ability and willingness of subject to give written informed consent.

Part I (vaccination phase) Exclusion Criteria:

1. Active infection with schistosomiasis or Treponema pallidum (syphilis).
2. Seropositive for VSV-G antibody, hepatitis B surface antigen (HBsAg) or concurrent chronic active hepatitis C.
3. Autoimmune diseases or clinically serious cardiac, pulmonary, gastrointestinal, hepatic, renal or neurologic disease, which in the opinion of the investigator will compromise ability to participate in the study.
4. Receipt of immune globulin or blood products within 90 days prior to study entry.
5. Receipt of any vaccinations within 30 days prior to study entry.
6. Previous receipt of any HIV vaccine. NOTE: Subjects who participated previously in an HIV vaccine trial who have documentation of receipt of only placebo may be eligible after discussion with the protocol chair.
7. Pregnancy and breast-feeding.
8. Prior systemic cancer chemotherapy,
9. Investigational agents and immunomodulators (cyclosporine, hematological growth factors, systemic corticosteroids, interleukins or interferons) within 90 days prior to study entry.

   NOTE: Subjects may be on antiretroviral agents not yet approved by the FDA as part of a clinical trial or expanded access program.
10. Anaphylaxis or allergy to vaccine components (See section 5.1.1).
11. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
12. Serious illness requiring systemic treatment and/or hospitalization until subject either completes therapy or is clinically stable on therapy, in the opinion of the investigator, for at least 30 days prior to study entry.
13. History of any AIDS-defining illness. NOTE: Subjects whose sole AIDS-defining illness is Kaposi's sarcoma limited to the skin that is not anticipated to require systemic therapy may be eligible after discussion with the protocol chair.
14. Nadir CD4 cell count <250 cell/mm3.
15. Changes in antiretroviral therapy for virologic failure prior to study entry.
16. Prisoners.

Part II (treatment interruption phase) Inclusion Criteria (Arm I and III only):

1. Receipt of three vaccinations . At the completion of the first 24 weeks of the study, potential eligible subjects for Part II will be unblinded, as to the receipt of active vaccine.

   NOTE: Subjects in Arm II and IV (vaccine placebo recipients) participation in the study will end with Part I.
2. Willingness to interrupt potent antiretroviral therapy for 12 weeks.
3. CD4 cell count > 500 cells/mm3 within 14 days prior to antiretroviral treatment interruption.

Part II Exclusion Criteria:

1. Confirmed viral flare, defined as two consecutive plasma HIV-1 RNA >5,000 copies/ml, during the immunization phase (Part I).
2. Development of any condition during the immunization phase that in the opinion of the investigator would place the subject at an increased risk for HIV viral rebound.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-09; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
• To evaluate the safety of a replication-defective HIV-1 vaccine (HIVAX™) in HIV-1 infected subjects on highly active antiretroviral therapy. | 48 weeks
  Frequency and severity of adverse events, laboratory abnormalities, and local and systemic reactogenicity signs and symptoms following vaccinations.
• To evaluate the potential immunogenicity of a replication-defective HIV-1 vaccine (HIVAX™) as determined by IFN-γ and IL-2 ELISPOT to pooled gag and env HIV peptides. | 48 weeks
  Magnitude of IFN-γ & IL-2 producing CD4+ and CD8+ T cells to pooled gag and env HIV peptides at 4 weeks post vaccinations.

SECONDARY OUTCOMES:
To explore the potential effectiveness of a replication-defective HIV-1 vaccine as a therapeutic vaccine | 48 weeks
  * Changes in CD4+ and CD8+ T-cell counts between the vaccine and placebo groups.
  * Changes in functional and phenotypic specific HIV gag and env induced T cell responses including in CD8 and CD4 T subsets.
  * HIV-1 RNA viral set point following antiretroviral treatment interruption, defined as the average of HIV-1 RNA values during the last two study visits of the antiretroviral treatment interruption.
  * Time to virologic rebound (HIV-1 RNA ≥ 5,000 copies/ml).
  * Breadth of HV-1 specific CD8+ T cell responses as determined by IFN-γ ELISPOT using overlapping HIV peptides for gag and env.
To monitor the impact of antiretroviral treatment interruption on viral resistance among subjects with virologic rebound (HIV-1 RNA ≥5,000 copies/ml) following resumption of antiretroviral treatment. | 16 weeks
  Treatment interruption: the number and percentage: 1)meet HIV-1 RNA (>2.0 fold above nadir and >5,000 copies/mL on two consecutive measurements verified at least one week apart) and CD4+ criteria (<400 cell/mm3 or 50% decreases from baseline in CD4 cell count on two consecutive measurements verified at least one week apart) to re-institute treatment before 12 wks; 2)genotypic resistance in re-emergent virus. Treatment resumption: the number and percentage: 1)meet criteria for virologic failure; 2)genotypic resistance in patients with virologic failure.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Fischl, MD, Study Director — University of Miami
Locations (1):
- University of Miami School of Medicine, AIDS Clinical Research unit, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pallikkuth S, Bolivar H, Fletcher MA, Babic DZ, De Armas LR, Gupta S, Termini JM, Arheart KL, Stevenson M, Tung FY, Fischl MA, Pahwa S, Stone GW. A therapeutic HIV-1 vaccine reduces markers of systemic immune activation and latent infection in patients under highly active antiretroviral therapy. Vaccine. 2020 Jun 2;38(27):4336-4345. doi: 10.1016/j.vaccine.2020.04.015. Epub 2020 May 6. PMID 32387010
- [Derived] Tung FY, Tung JK, Pallikkuth S, Pahwa S, Fischl MA. A therapeutic HIV-1 vaccine enhances anti-HIV-1 immune responses in patients under highly active antiretroviral therapy. Vaccine. 2016 Apr 27;34(19):2225-32. doi: 10.1016/j.vaccine.2016.03.021. Epub 2016 Mar 19. PMID 27002500